CLINICAL TRIAL: NCT01102647
Title: Assessment of Cholesterol Metabolism in Heterozygous Phytosterolemia
Brief Title: Cholesterol Metabolism in Heterozygous Phytosterolemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Peter J Jones, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B2009:133
Record Dates: First submitted 2010-04-07; First posted 2010-04-13 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phytosterol ester (Experimental): Plant sterol compared with placebo
  Interventions: Dietary Supplement: phytosterol ester

INTERVENTIONS:
Dietary Supplement: phytosterol ester — 1.6 g phytosterols/day for 29 days
  Other Names: Phytocell Phytosterols, NPN#: 80012048

SUMMARY:
The purpose of the study is to examine the effect of plant sterols on cholesterol absorption and synthesis in people with heterozygous phytosterolemia.

DETAILED DESCRIPTION:
A plant sterol supplementation study will be conducted in individuals who are heterozygous for phytosterolemia compared to non-carriers. The study will use a double-blind, randomised, crossover, placebo-controlled design in which participants will consume 2 treatments including 1.6 g of plant sterol pills and a placebo pill, each for 4 weeks. A 4 week washout period will separate the two treatment periods. Plant sterol concentrations will be measured by gas liquid chromatography and absorption will be measured by the ratio of campesterol to lathosterol in plasma. Cholesterol absorption and synthesis will be measured by dual stable isotope technique, involving simultaneous administration of 13C-cholesterol and deuterium oxide, respectively.

ELIGIBILITY:
Inclusion Criteria:

* heterozygous for phytosterolemia, wild-type.

Exclusion Criteria:

* Pregnant,
* Previous heart attack,
* Kidney disease.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Decrease in plasma LDL-cholesterol | 29 days
  Other studies have found 10% reduction in plasma LDL-cholesterol after 2.2-3.2 gram of plant sterol supplementation for 4 weeks in heterozygous phytosterolemia.

SECONDARY OUTCOMES:
Increase plasma plant sterols | 29 days
  We will use a control group and compare the level of increase in plasma plant sterol levels in both group over the course of plant sterol consumption

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Jones, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Myrie SB, Mymin D, Triggs-Raine B, Jones PJ. Serum lipids, plant sterols, and cholesterol kinetic responses to plant sterol supplementation in phytosterolemia heterozygotes and control individuals. Am J Clin Nutr. 2012 Apr;95(4):837-44. doi: 10.3945/ajcn.111.028985. Epub 2012 Feb 29. PMID 22378727